CLINICAL TRIAL: NCT01155999
Title: Clinical Efficacy and Safety of T1225 Versus Tobramycin 0.3 % Eye Drops in the Treatment of Purulent Bacterial Conjunctivitis of Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT1225-PIIIB-02/08; 2008-003567-39 (EudraCT Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2011-09

CONDITIONS: Purulent Bacterial Conjunctivitis
MeSH Terms: interventions — Tobramycin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- T1225 (Experimental)
  Interventions: Drug: T1225
- Tobramycin (Active Comparator)
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: T1225 — one drop twice daily (morning and evening) in each eye from Day 0 to Day 2
  Arms: T1225
Drug: Tobramycin — 1 to 2 drops every two hours while awake on Days 0-1, up to 8×/day, then 1 to 2 drops 4 times daily on Days 2-6
  Arms: Tobramycin

SUMMARY:
Efficacy/Safety of T1225, in comparison to reference product, for the treatment of purulent bacterial conjunctivitis of children.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ one day of life and ≤ 18 years
* Purulent bacterial conjunctivitis

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 286 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T1225 | Tobramycin
Started | 146 | 140
Completed | 139 | 136
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T1225 | Tobramycin | Total
Number analyzed (Participants) | 146 | 136 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.06 (3.40) | 3.52 (4.17) | 3.28 (3.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 68 | 144
  Male | 70 | 68 | 138
Region of Enrollment [Number; unit: participants]
  France | 15 | 11 | 26
  Germany | 14 | 11 | 25
  Italy | 2 | 2 | 4
  Poland | 19 | 17 | 36
  Portugal | 2 | 4 | 6
  Romania | 29 | 28 | 57
  Algeria | 18 | 17 | 35
  Tunisia | 47 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Variable Was Clinical Cure in the Worse Eye on Day 3
Description: Clinical cure was defined as a score 0 for bulbar conjunctival injection (evaluated using a 4 point ordinal scale) and a score 0 for conjunctival purulent discharge (evaluated using a 4 point ordinal scale).
Time Frame: Day 3
Population: The analysis of the primary clinical efficacy variable was primarily performed on the basis of the MFAS. The MFAS consisted of all patients of the FAS with positive Day 0 culture results in an eligible eye.
Measure: Number; unit: participants
Arm/Group | T1225 | Tobramycin
Number analyzed (Participants) | 102 | 101
participants | 48 | 29

ADVERSE EVENTS:
Arm/Group | T1225 | Tobramycin
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/140
Other Adverse Events (participants affected / at risk) | 0/146 | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.